CLINICAL TRIAL: NCT05477862
Title: Neural Mechanisms of Induced Calmness After Listening to Improvisatory Music: An Investigation for Healthy Individuals and Persons With Alzheimer's Dementia
Brief Title: Neural Mechanisms of Clinically Designed Improvisatory Music for Alzheimer's Disease
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Northwestern University (Other)
Responsible Party: Principal Investigator, Borna Bonakdarpour, Associate Professor of Neurology, Northwestern University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 00215983
Record Dates: First submitted 2022-07-17; First posted 2022-07-28 (Actual); Last update posted 2024-03-22 (Actual); Status verified 2024-03

CONDITIONS: Alzheimer Disease
Keywords: Anxiety; Alzheimer; Dementia; Agitation; Irritability; Music Intervention; Music Medicine; Music Improvisation
MeSH Terms: conditions — Alzheimer Disease; Anxiety Disorders; Dementia; Psychomotor Agitation

STUDY DESIGN:
Intervention Model Description: 15 individuals with Alzheimer Disease (AD) and 15 cognitively healthy individuals.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Alzheimer Disease (AD) (Experimental)
  Interventions: Behavioral: Clinically Designed Improvisatory Music
- Cognitively Healthy (CH) (Experimental)
  Interventions: Behavioral: Clinically Designed Improvisatory Music

INTERVENTIONS:
Behavioral: Clinically Designed Improvisatory Music — Clinically Designed Improvisatory Music (CDIM) is a form of improvised music based on calm-inducing sound parameters which brought relief to our cohort of neurology patients.

SUMMARY:
Clinically Designed Improvisatory Music (CDIM) is a form of improvised music based on calm-inducing sound parameters which brought relief to our cohort of neurology patients. As a direct sound-based approach, CDIM does not rely on autobiographical memory and may have wider applicability and generalizability. We wish to examine if CDIM decreases anxiety in 15 cognitively healthy individuals and 15 Alzheimer Disease patients with anxiety (AD-A).

DETAILED DESCRIPTION:
The goal of this study is to identify the neural mechanisms of induced calmness through live clinically designed improvisatory music (CDIM) in cognitively healthy individuals and persons with Alzheimer's dementia suffering from agitation. This study is novel as most music interventions for dementia use familiar music and the underlying neural mechanism of calmness induced by music is not well known. We plan to investigate changes in 3 major large-scale brain networks using functional magnetic resonance imaging (fMRI). The major questions we plan to answer are as follows: 1. How does improvisatory music change the connectivity within brain emotion related networks in neurotypical individuals? 2. Does improvisatory music induce a state of calmness in individuals with Alzheimer's dementia and how? Based on objective evidence provided by this study we can justify further usage of music for patients with Alzheimer's, in particular, in the form of improvisation.

ELIGIBILITY:
Inclusion Criteria:

1. Cognitively healthy individuals

   Cognitively healthy control participants evaluated through the Northwestern Mesulam Center. BAI > 8.

   Exclusion Criteria: hearing loss
2. Individuals with mild to moderate Alzheimer's disease

This group will similarly be recruited through the Mesulam Center. All individuals recruited by the research Core at the center are well characterized tests standardized across all NIH funded Alzheimer Centers across the nation. Individuals with mild to moderate neurocognitive disorder due to AD will have an MMSE greater than >15 and Clinical Dementia Rating (CDR) between 0.5 and 2.. They will also have a history of neurocognitive-related agitation/anxiety, and a Beck Anxiety Index (BAI) greater than 8, suggestive of at least a mild level of anxiety.

Exclusion criteria: MMSE<15, CDR>2, hearing loss

Ages: 55 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2023-10-15 (Actual); Primary Completion 2025-10-15 (Estimated); Study Completion 2026-01-15 (Estimated)

PRIMARY OUTCOMES:
Change in Neuropsychiatric Inventory (NPI) [NPI-1: pre-intervention; NPI-2: post-intervention] | Through study completion (3 years)
  Change in NPI (NPI-2 minus NPI-1)
Change in Beck Anxiety Inventory [BAI-1: pre-intervention; BAI-2: post-intervention] | Through study completion (3 years)
  Change in BAI (BAI-2 minus BAI-1)

SECONDARY OUTCOMES:
Change in Systolic Blood Pressure [SBP-1: pre-intervention; SBP-2: post-intervention] | Through study completion (3 years)
  Change in SBP (SBP-2 minus SBP-1)
Change in Heart rate [HR-1: pre-intervention; HR-2: post-intervention] | Through study completion (3 years)
  Change in HR (HR-2 minus HR-1)
Change Respiratory Rate [RR-1: pre-intervention; RR-2: post-intervention] | Through study completion (3 years)
  Change in RR (RR-2 minus RR-1)
Change in Skin conductance [SC-1: pre-intervention; SC-2: post-intervention] | Through study completion (3 years)
  Change in SC (SC-2 minus SC-1)
Change in Resting state functional connectivity MRI | Through study completion (3 years)
  Functional Connectivity within three resting state networks: Change in Default Network (DN), Change in Salience Network (SN), and Change in Reward Network (RN).

CONTACTS AND LOCATIONS:
Overall Officials: Borna Bonakdarpour, MD, FAAN, Principal Investigator — Northwestern Mesulam Center for Cognitive Neurology and Alzheimer Disease
Locations (1):
- Mesulam Center for Cognitive Neurology and Alzheimer's Disease, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Bonakdarpour B, McFadden A, Zlotkowski S, Huang D, Shaker M, Shibata B, Haben W, Brashear C, Sandoval A, Breitenbach C, Rodriguez C, Viamille J, Porter M, Galic K, Schaeve M, Thatcher D, Takarabe C. Neurology Telemusic Program at the Time of the COVID-19 Pandemic: Turning Hospital Time Into Aesthetic Time During Crisis. Front Neurol. 2021 Dec 13;12:749782. doi: 10.3389/fneur.2021.749782. eCollection 2021. PMID 34966344
- [Background] Lyketsos CG, Carrillo MC, Ryan JM, Khachaturian AS, Trzepacz P, Amatniek J, Cedarbaum J, Brashear R, Miller DS. Neuropsychiatric symptoms in Alzheimer's disease. Alzheimers Dement. 2011 Sep;7(5):532-9. doi: 10.1016/j.jalz.2011.05.2410. PMID 21889116
- [Background] Baird A, Samson S. Music and dementia. Prog Brain Res. 2015;217:207-35. doi: 10.1016/bs.pbr.2014.11.028. Epub 2015 Jan 31. PMID 25725917
- [Background] Assal F, Cummings JL. Neuropsychiatric symptoms in the dementias. Curr Opin Neurol. 2002 Aug;15(4):445-50. doi: 10.1097/00019052-200208000-00007. PMID 12151841
- [Background] Seeley WW, Menon V, Schatzberg AF, Keller J, Glover GH, Kenna H, Reiss AL, Greicius MD. Dissociable intrinsic connectivity networks for salience processing and executive control. J Neurosci. 2007 Feb 28;27(9):2349-56. doi: 10.1523/JNEUROSCI.5587-06.2007. PMID 17329432